CLINICAL TRIAL: NCT02274116
Title: Repetitive Exposure of Intermittent Hypoxia to Enhance Walking Recovery in Persons With Chronic Spinal Cord Injury
Brief Title: Acute Intermittent Hypoxia on Leg Function Following Spinal Cord Injury
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Foundation Wings For Life (Other)
Responsible Party: Principal Investigator, Randy Trumbower, PT, PhD, Assistant Professor, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017P001940c
Record Dates: First submitted 2014-10-06; First posted 2014-10-24 (Estimated); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injuries
Keywords: acute intermittent hypoxia; walking; spasticity; incomplete spinal cord injury; breathing; strength
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Hypoxia (AIH) (Active Comparator): Subjects with chronic, motor-incomplete SCI will breath mild bouts of low oxygen.
  Intervention: AIH - Intermittent Hypoxia - hypoxia air mixture Dosage: 10% oxygen Frequency: 1.5 minutes bouts of low oxygen with 1.0 minute intervals of room air Duration: 38 minutes
  Interventions: Other: AIH - Intermittent Hypoxia - hypoxia air mixture
- Intermittent Room Air (SHAM) (Sham Comparator): Subjects with chronic, motor-incomplete SCI will breath mild bouts of room air.
  Intervention: SHAM - Intermittent Room Air - room air mixture Dosage: 21% oxygen Frequency: 1.5 minutes bouts of room air with 1.0 minute intervals also of room air Duration: 38 minutes
  Interventions: Other: SHAM - Intermittent Room Air - room air mixture

INTERVENTIONS:
Other: SHAM - Intermittent Room Air - room air mixture — Participants will breathe intermittent room air via air generators. The generators will fill reservoir bags attached to a non-rebreathing face mask. Oxygen concentration will be continuously monitored to ensure delivery of fraction of inspired oxygen (FIO2)=0.21±0.02 (normoxia). Participants will receive treatment 5 times per week for 2 weeks.
  Arms: Intermittent Room Air (SHAM)
Other: AIH - Intermittent Hypoxia - hypoxia air mixture — Participants will breathe intermittent low oxygen via air generators. The generators will fill reservoir bags attached to a non-rebreathing face mask. Oxygen concentration will be continuously monitored to ensure delivery of fraction of inspired oxygen (FIO2)=0.10±0.02 (hypoxia). Participants will receive treatment 5 times per week for 2 weeks.
  Arms: Intermittent Hypoxia (AIH)

SUMMARY:
The purpose of this study is to determine how the nervous system controlling leg muscles is altered following spinal cord injury and how they may be affected by brief periods of low oxygen inhalation over time.

The investigators hypothesize:

* Acute intermittent hypoxia (AIH) exposure will increase maximum voluntary leg strength in persons with incomplete cervical spinal cord injury (SCI)
* AIH exposure will increase multijoint reflex excitability of leg muscles in persons with incomplete cervical SCI
* AIH exposure will increase walking performance in persons with incomplete cervical SCI

DETAILED DESCRIPTION:
Accumulating evidence suggests that repeatedly breathing low oxygen levels for brief periods (termed intermittent hypoxia) is a safe and effective treatment strategy to promote meaningful functional recovery in persons with chronic spinal cord injury. Repetitive exposure to mild hypoxia triggers a cascade of events in the spinal cord, including new protein synthesis and increased sensitivity in the circuitry necessary for breathing and walking. Recently, the investigators demonstrated that daily (5 consecutive days) of intermittent hypoxia stimulated walking enhancement in persons with chronic spinal cord injury.

Despite these exciting findings, important clinical questions remain. For example, the investigators do not know if prolonged, but less intense intermittent hypoxia induces longer-lasting motor recovery as has been shown in rat models. The investigators hypothesize that repetitive exposures to modest bouts of low oxygen will enhance and prolong walking recovery in persons with chronic spinal cord injury. The investigators anticipate intermittent hypoxia-induced improvements in overground walking ability, likely due to greater balance in excitatory and inhibitory neural transmission. Whereas excitatory inputs drive walking, inhibitory inputs sculpt and coordinate muscle activity; yet so often remain compromised after chronic injury. Thus, the investigators also predict that repetitive exposures to intermittent hypoxia will result in improved inhibition and subsequently enhance muscle coordination during walking. The investigators will use multiple experimental approaches, including muscle electromyography, measurements of walking dynamics and stretch reflexes. Finally, it is critical to assure that repetitive exposures to intermittent hypoxia do not elicit pathologies characteristic of more severe, chronic hypoxia experienced by individuals with obstructive sleep apnea. The investigators will confirm that repetitive exposure to mild bouts of intermittent hypoxia is safe.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old (the latter to reduce likelihood of heart disease);
* medically stable with clearance from physician to participate;
* motor---incomplete SCI at C2---L5 with non---progressive etiology;
* >6 months since SCI to ensure minimal confounds of spontaneous neurological recovery;
* those classified as ambulatory must have the ability to advance one step overground without human assistance.

Exclusion Criteria:

* concurrent illness, including unhealed decubiti, severe neuropathic or chronic pain syndrome, infection, cardiovascular disease, osteoporosis (history of fractures), active heterotopic ossification, or known history of peripheral nerve injury to legs;
* less than 24 on the Mini-mental Exam;
* recurrent autonomic dysreflexia
* cardiopulmonary complications
* concurrent physical therapy
* pregnancy because of unknown effects of AIH on a fetus, although women will not otherwise be excluded

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-10; Primary Completion 2027-08 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in overground walking endurance | Baseline, immediately following intervention (day 5), and at 1, 2, and 4 weeks
  walking endurance (6 minute walk test - how far one can walk in 6 minutes)

SECONDARY OUTCOMES:
Change in overground walking speed | Baseline, immediately following intervention (day 5), and at 1, 2, and 4 weeks
  walking speed (10 meter walk test - how fast one can walk in 10 meters)

CONTACTS AND LOCATIONS:
Overall Officials: Randy D Trumbower, PT, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Cambridge, Massachusetts, United States

REFERENCES:
- [Background] Hayes HB, Jayaraman A, Herrmann M, Mitchell GS, Rymer WZ, Trumbower RD. Daily intermittent hypoxia enhances walking after chronic spinal cord injury: a randomized trial. Neurology. 2014 Jan 14;82(2):104-13. doi: 10.1212/01.WNL.0000437416.34298.43. Epub 2013 Nov 27. PMID 24285617
- [Background] Trumbower RD, Jayaraman A, Mitchell GS, Rymer WZ. Exposure to acute intermittent hypoxia augments somatic motor function in humans with incomplete spinal cord injury. Neurorehabil Neural Repair. 2012 Feb;26(2):163-72. doi: 10.1177/1545968311412055. Epub 2011 Aug 5. PMID 21821826
- [Background] Lovett-Barr MR, Satriotomo I, Muir GD, Wilkerson JE, Hoffman MS, Vinit S, Mitchell GS. Repetitive intermittent hypoxia induces respiratory and somatic motor recovery after chronic cervical spinal injury. J Neurosci. 2012 Mar 14;32(11):3591-600. doi: 10.1523/JNEUROSCI.2908-11.2012. PMID 22423083
- [Background] Dale-Nagle EA, Hoffman MS, MacFarlane PM, Satriotomo I, Lovett-Barr MR, Vinit S, Mitchell GS. Spinal plasticity following intermittent hypoxia: implications for spinal injury. Ann N Y Acad Sci. 2010 Jun;1198:252-9. doi: 10.1111/j.1749-6632.2010.05499.x. PMID 20536940